CLINICAL TRIAL: NCT00002060
Title: A Multi-Center Randomized Double-Blind Placebo-Controlled Study To Investigate the Effect of Isoprinosine in Patients With AIDS Related Complex (ARC)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Newport Pharmaceuticals International (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Masking: Double | Purpose: Treatment
Other Study IDs: 008D; ISO-111-USA
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1989-06

CONDITIONS: HIV Infections
Keywords: AIDS-Related Opportunistic Infections; Inosine Pranobex; Homosexuality; Acquired Immunodeficiency Syndrome; AIDS-Related Complex
MeSH Terms: conditions — HIV Infections; AIDS-Related Opportunistic Infections; Homosexuality; Acquired Immunodeficiency Syndrome; AIDS-Related Complex | interventions — Inosine Pranobex

INTERVENTIONS:
Drug: Inosine pranobex

SUMMARY:
The objective is to determine the effect of Isoprinosine (inosine pranobex) in homosexual male patients with AIDS related complex (ARC) in delaying the onset of AIDS. Secondly, to determine the effect of Isoprinosine in decreasing the severity and/or incidence of lesser opportunistic infections and/or other conditions associated with ARC.

ELIGIBILITY:
Exclusion Criteria

Concurrent Medication:

Excluded:

* Cardiac glycosides.

Patients with the following are excluded:

* AIDS.
* Presenting with chronic candida infection-colo/rectal, oral/pharyngeal, cutaneous (finger/toenails) - for = or > 3 months who have not responded to therapy.
* Critical illness.
* Hemophilia.

Prior Medication:

Excluded within 1 month of study entry:

* Steroids.
* Cytotoxic immunosuppressive agents.
* Radiotherapy and/or systemic antiviral medication.
* Immunomodulators (including Isoprinosine).

Prior Treatment:

Excluded within 1 month of study entry:

* Radiotherapy.

History of gout, uric acid urolithiasis, uric acid nephrolithiasis, or renal dysfunction.

* Lymphoid malignancy.

Homosexual male patients with AIDS related complex (ARC).

Current IV drug abuse.

Ages: 18 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (1):
- Newport Pharmaceuticals International Inc, Laguna Hills, California, United States